CLINICAL TRIAL: NCT07348848
Title: Prospective Evaluation of Foreign Body Airway Obstruction Interventions Among Infants: A Non-randomized Pilot Cohort Study
Brief Title: Prospective Evaluation of Foreign Body Airway Obstruction Interventions Among Infants
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Cody Dunne, Primary Investigator, Emergency Physician, University of Calgary
Other Study IDs: REB25-0419B
Record Dates: First submitted 2025-09-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Foreign Body Airway Obstruction
Keywords: Choking; Infants; Prospective cohort; Feasibility
MeSH Terms: conditions — Airway Obstruction | interventions — Heimlich Maneuver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants with FBAO: Infants (aged 2 years or younger) with a foreign body airway obstruction who are conscious when they receive their first intervention
  Interventions: Procedure: Chest compressions/thrusts; Procedure: Back blows; Procedure: Abdominal Thrusts

INTERVENTIONS:
Procedure: Chest compressions/thrusts — Chest compressions or thrusts received as first intervention
Procedure: Back blows — Back blows received as first intervention
Procedure: Abdominal Thrusts — Abdominal thrusts received as first intervention

SUMMARY:
Foreign body airway obstruction (FBAO, choking) is a life-threatening emergency requiring time-sensitive treatment to prevent severe injury or deaths. Traditional treatments taught in first aid courses include abdominal thrusts, back blows, and chest compressions or thrusts. Currently, first aid guidelines recommend different treatments for adults, child and infants.

Until recently, data on these techniques was limited to case series from the late 1900's. To further improve our knowledge of which treatment is most effective and safest for patients, this study will collect data on choking incidents in Alberta, Canada. The first phase of this project will make sure identifying and recruiting choking patients in real-time is possible so that the highest quality of data can be collected. If successful, this study will support a future project where the different choking treatments are compared in terms of their effectiveness and safety. This study will focus on infants aged 2 years or younger.

ELIGIBILITY:
Inclusion Criteria:

* Infants (aged 2 years or less) who experienced an out-of-hospital FBAO in Alberta, Canada
* Received a FBAO intervention while conscious by bystander or healthcare provider
* Were assessed by EMS at the time of the incident, or later attended an emergency department due to the incident

Exclusion Criteria:

* Patients with abnormal airway anatomy such as a tracheostomy.
* Patients who were unconscious when they received the initial FBAO intervention

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants (aged 2 years or less) who experienced an out-of-hospital FBAO and received a FBAO intervention while conscious in Alberta, Canada, and, subsequently, were assessed by EMS or at an emergency department
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Eligible patient recruitment | Through study completion, a 6 month period
  Count of eligible patients recruited per month

SECONDARY OUTCOMES:
Proportion of eligible patients recruited | Through study completion, a 6 month period
  Among patients who screen as eligible for recruitment, the proportion of those who are successfully recruited
Proportion of recruited patients with satisfactory data collection | Through study completion, a 6 month period
  Among patients successfully recruited, the those patients with >= 90% of desired variables collected
Foreign body airway obstruction relief | Day 1
  Defined as: responders determining that the patient did not require further FBAO intervention due to improvement or resolution of their respiratory distress in a conscious patient, or the ability for a responder to successfully ventilate an unconscious patient when previously they were unable to due to obstruction
Survival to acute care discharge | From date of enrolment until the date of acute care discharge or date of death from any cause, whichever came first, assessed up to 3 month
  Defined as discharge from the care of Emergency Medical Services(EMS) or paramedics, the emergency department, or the hospital.
Survival to acute care discharge with favourable neurological outcome | From date of enrolment until the date of acute care discharge or date of death from any cause, whichever came first, assessed up to 3 month
  Defined as the patient being able to be discharge to the home environment that they previously lived, with the ability to perform the same activities of daily living as before the FBAO incident
Intervention-associated injuries | From date of enrolment until the date of acute care discharge or date of death from any cause, whichever came first, assessed up to 3 month
  Listed summary of any injuries reported among patient recruited for study occurring as a result of the FBAO intervention as determined by the treating physician/care provider

CONTACTS AND LOCATIONS:
Locations (1):
- Virtual, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT07348848/Prot_SAP_000.pdf